CLINICAL TRIAL: NCT06508359
Title: Prophylactic vs Rescue Norepinephrine and Phenylephrine for Spinal Anesthesia-induced Hypotension on Neonatal Outcomes During Cesarean Section: A Multicenter, Single-blind, Crossover, Factorial Cluster Trial
Brief Title: Norepinephrine and Phenylephrine for Spinal Anesthesia-induced Hypotension.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2025-1
Record Dates: First submitted 2024-07-14; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Outcome
Keywords: Spinal anesthesia-induced hypotension; Norepinephrine; Phenylephrine; Neonatal outcomes; Cesarean section
MeSH Terms: interventions — Norepinephrine; Vasoconstrictor Agents; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prophylactic norepinephrine group (Experimental): A maintenance dose of norepinephrine (0.05 ug/kg/min) infusion simultaneous with spinal anesthesia. The maternal systolic blood pressure was consistently maintained above 80% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery.
  Interventions: Drug: Norepinephrine
- Prophylactic phenylephrine group (Experimental): A maintenance dose of phenylephrine (0.625 ug/kg/min) infusion simultaneous with spinal anesthesia. The maternal systolic blood pressure was consistently maintained above 80% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery.
  Interventions: Drug: Phenylephrine
- Rescue norepinephrine group (Active Comparator): The maternal systolic blood pressure was consistently maintained above 80% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery. Spinal anesthesia-induced hypotension is managed by administering a 6 μg intravenous bolus of norepinephrine.
  Interventions: Drug: Norepinephrine
- Rescue phenylephrine group (Active Comparator): The maternal systolic blood pressure was consistently maintained above 80% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery. Spinal anesthesia-induced hypotension is managed by administering a 75 μg intravenous bolus of phenylephrine.
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Norepinephrine — Prophylactic or rescue norepinephrine for spinal anesthesia-induced hypotension
  Other Names: Vasopressor
  Arms: Prophylactic norepinephrine group; Rescue norepinephrine group
Drug: Phenylephrine — Prophylactic or rescue phenylephrine for spinal anesthesia-induced hypotension
  Other Names: Vasopressor
  Arms: Prophylactic phenylephrine group; Rescue phenylephrine group

SUMMARY:
This study aims to explore the effects of different application modes (prophylactic and rescue strategy) of norepinephrine and norepinephrine on neonate umbilical artery pH undergoing cesarean section.

DETAILED DESCRIPTION:
Spinal anesthesia-induced hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of spinal anesthesia-induced hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. The 2016 ASA guidelines for obstetric anesthesia suggest avoiding hypotension following spinal anesthesia in women and emphasize the use of vasopressors, specifically alpha-receptor agonists, as the preferred strategy to prevent and manage spinal anesthesia-induced hypotension. The prophylactic vasopressor strategy is more effective in enhancing hemodynamic stability and reducing adverse events such as nausea and vomiting during cesarean section, compared to rescue strategy. However, it does not demonstrate significant advantages in neonatal outcomes such as umbilical artery pH and Apgar score. The impact of various vasopressor application patterns on neonatal outcomes after cesarean section lacks further supporting evidence. Therefore, this study aims to explore the effects of different application modes (prophylactic and rescue strategy) of norepinephrine and norepinephrine on neonate umbilical artery pH undergoing cesarean section through a multicenter, single-blind, 2*2 crossover and cluster randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥37 weeks
* American Society of Anesthesiologists physical status classification II
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥140 mmHg
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
pH | Immediately after delivery
  From umbilical arterial blood gases.
Base excess (BE) | Immediately after delivery
  From umbilical arterial blood gases.

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline
The incidence of bradycardia | 1-15 minutes after spinal anesthesia
  Heart rate < 60 beats/min
The incidence of nausea and vomiting | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline.
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University